CLINICAL TRIAL: NCT02461693
Title: Evaluating the Role of Expectations in Response to Caffeine Consumption: A Randomized Control Trial
Brief Title: Evaluating the Role of Expectations in Response to Caffeine Consumption: An RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Allison, Phd, Associate Dean for Science, School of Public Health, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: F150410009
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Caffeine; Affect; Cognitive Ability, General; Mood
Keywords: Vigilance; Mood; Randomized Controlled Trial; Probability
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants, study personnel interacting with participants, and investigators were blinded. Only the study statistician knew treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine (Experimental): One-time treatment with 200mg caffeine pill
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): One-time treatment with lactose-based placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine — 200mg delivered as pill; one-time dose
  Arms: Caffeine
Drug: Placebo — Lactose-based pill; one-time dose
  Arms: Placebo

SUMMARY:
The purpose of this project is to examine the effect of expectancy on mood and alertness after consumption of caffeine "treatment" or placebo "control" pill, given that participants know their probability for receiving the caffeine versus placebo pill. Participants will be randomly assigned a probability (ranging from 0-100%) of receiving caffeine vs. placebo, and this probability will be revealed to them before consumption of the assigned pill and subsequent cognitive testing. At the time of consumption, neither study staff administering the intervention nor participants will know for certain which pill is given to each participant. Pill assignment will depend on pre-determined randomization probabilities, which will be provided and assigned by the study statistician. By revealing participants' individual probability of receiving the caffeine pill, we will induce positive or negative expectancies regarding likelihood for receipt of the caffeine pill. These experimental manipulations will: 1) estimate the effect of expectancy on cognitive and affective outcomes, and 2) allow for a more direct estimate of the effect of the caffeine pill under real-world conditions than would a conventional randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years-old or older
* available to participate on the dates specified
* willing to take a caffeine or placebo pills at study session
* willingness to abstain from caffeine for 12 hours prior to study visit (8:30pm-8:30am)
* UAB employees or students with some college education (including current enrollment)

Exclusion Criteria:

* self-reported use of ADHD medication
* self-reported use of anxiety medication
* self-reported use of sleep medication
* self-reported use of nicotine products
* self-reported lactose intolerance
* self-reported uncorrected vision
* self-reported pregnancy or trying to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B Allison, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Raw de-identified data will be posted as a replication data set on ICPSR after publication of results in a journal. Data will be free to download and accessible to anyone with access to ICPSR replication data sets.

REFERENCES:
- [Result] George BJ, Li P, Lieberman HR, Pavela G, Brown AW, Fontaine KR, Jeansonne MM, Dutton GR, Idigo AJ, Parman MA, Rubin DB, Allison DB. Randomization to randomization probability: Estimating treatment effects under actual conditions of use. Psychol Methods. 2018 Jun;23(2):337-350. doi: 10.1037/met0000138. Epub 2017 Apr 13. PMID 28406674

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: One-time treatment with lactose-based placebo pill
  Placebo
Period: Overall Study
Arm/Group | Caffeine | Placebo
Started | 103 | 102
Completed | 103 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caffeine | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 5 participants (3 assigned to caffeine and two assigned to placebo) were deemed ineligible for study after participation and were thus excluded from the analysis
  years | 33.83 (14.02) | 29.75 (11.39) | 31.79 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5 participants (3 assigned to caffeine and two assigned to placebo) were deemed ineligible for study after participation and were thus excluded from the analysis
  Participants
    Female | 62 | 61 | 123
    Male | 38 | 39 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 5 participants (3 assigned to caffeine and two assigned to placebo) were deemed ineligible for study after participation and were thus excluded from the analysis
  Participants
    Hispanic or Latino | 1 | 7 | 8
    Not Hispanic or Latino | 84 | 75 | 159
    Unknown or Not Reported | 15 | 18 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 5 participants (3 assigned to caffeine and two assigned to placebo) were deemed ineligible for study after participation and were thus excluded from the analysis
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 16 | 12 | 28
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 39 | 50 | 89
    White | 39 | 30 | 69
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Mood State Score on POMS-2 Test
Description: Profile of Mood States (POMS-2)- "Volunteers rated a series of 65 mood-related adjectives with regard to how they were feeling "right now" on a scale of 0 (not at all) to 4 (extremely). The adjectives factor into six mood sub-scales: Tension-Anxiety; Depression-Dejection; Anger-Hostility; Vigor-Activity; Fatigue-Inertia; Confusion-Bewilderment and a Total Mood Disturbance score which aggregates the six sub-scales into a single variable." - from our publication. The minimum and maximum possible raw scores were: 0 and 40 for Tension-Anxiety, 0 and 52 for Depression-Dejection, 0 and 44 for Anger-Hostility, 0 and 36 for Vigor-Aactivity, 0 and 24 for Fatigue-Inertia, 0 and 40 for Confusion-Bewilderment, -36 and 200 for Total Mood Disturbance, and 0 and 24 for Friendliness. For Friendliness and Vigor-Activity, the more positively a person feels, the higher the score. For all other sub-scales and Total Mood Disturbance, the more negatively a person feels, the higher the score.
Time Frame: 30 minutes post pill consumption
Population: Results are of raw data as presented in our publication
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 100 | 100
units on a scale
  Total Mood Displacement: number analyzed (Participants) | 88 | 89
  Total Mood Displacement | 2.63 (1.98) | 14.08 (2.86)
  Anger-Hostility: number analyzed (Participants) | 94 | 99
  Anger-Hostility | 2.19 (0.38) | 2.54 (0.46)
  Confusion-Bewilderment: number analyzed (Participants) | 99 | 99
  Confusion-Bewilderment | 6.23 (0.48) | 7.00 (0.53)
  Depression-Dejection: number analyzed (Participants) | 98 | 95
  Depression-Dejection | 1.87 (0.35) | 3.15 (0.61)
  Fatigue-Inertia: number analyzed (Participants) | 97 | 99
  Fatigue-Inertia | 4.44 (0.49) | 6.65 (0.68)
  Friendliness: number analyzed (Participants) | 99 | 100
  Friendliness | 13.47 (0.47) | 12.97 (0.44)
  Tension-Anxiety: number analyzed (Participants) | 98 | 97
  Tension-Anxiety | 5.53 (0.52) | 5.81 (0.52)
  Vigor-Activity: number analyzed (Participants) | 99 | 100
  Vigor-Activity | 16.35 (0.73) | 13.13 (0.69)

2. Primary Outcome: Vigilance Score on Computer-based Test Using Random, Visual Stimulus: Proportion Correct (Out of 60)
Description: Scanning Visual Vigilance Test. "This test assesses vigilance, ability to sustain attention during long, boring, continuous tasks that generate minimal cognitive load (Fine et al, 1994; Lieberman et al, 1998; 2002). The volunteer continuously scans a computer screen to detect an infrequent, difficult-to-detect stimulus that appears at random intervals and locations for 2 s. On average, a stimulus was presented once per minute. Upon detection of the stimulus, the volunteer pressed the space bar as rapidly as possible. Whether a stimulus was detected and time required for detection was recorded. Responses before or after stimulus occurrence were false alarms. The test lasted 60 minutes." - from our publication
Time Frame: 45 to 105 minutes post pill consumption
Population: One participant who received the caffeine pill had to use the restroom during the vigilance testing period and had to stop the test. Due to a technicality of the computer program, her data for the vigilance test was not available for analysis.
Measure: Mean (Standard Error); unit: Proportion correct
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 99 | 100
Proportion correct | 0.932 (0.014) | 0.888 (0.017)

3. Primary Outcome: Vigilance Score on Computer-based Test Using Random, Visual Stimulus: Number Correct, Number of False Alarm Hits
Description: as for outcome 2
Time Frame: 45 to 105 minutes post pill consumption
Population: as for outcome 2
Measure: Mean (Standard Error); unit: counts
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 99 | 100
counts
  Number correct (out of 60) | 55.9 (0.85) | 53.3 (1.00)
  Number of False Alarm Hits | 4.21 (0.67) | 5.80 (1.01)

4. Primary Outcome: Vigilance Score on Computer-based Test Using Random, Visual Stimulus: Mean Time to a Correct Hit
Description: as for outcome 2
Time Frame: 45 to 105 minutes post pill consumption
Population: as for outcome 2
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 99 | 100
seconds | 0.74 (0.03) | 0.88 (0.03)

ADVERSE EVENTS:
Time Frame: Three months
Description: No adverse events were reported
Arm/Group | Caffeine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/102
Other Adverse Events (participants affected / at risk) | 0/103 | 0/102

LIMITATIONS AND CAVEATS:
Please refer to our publication in Psyhcological Methods

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes